CLINICAL TRIAL: NCT00717171
Title: Efficacy of the SurgiStim3 Electrical Stimulation Device in Persons Undergoing Anterior Cruciate Ligament Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: VQ OrthoCare (Industry)
Responsible Party: Michelle Ocelnik, VQ OrthoCare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S060501-ACL
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Anterior Cruciate Ligament
Keywords: electrical stimulation; pain; medication; edema; interferential; neuromuscular; high voltage pulsed current; knee
MeSH Terms: conditions — Pain; Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Device: SurgiStim3
- 2 (Experimental)
  Interventions: Device: SurgiStim3

INTERVENTIONS:
Device: SurgiStim3 — Electrical stimulation device that provides interferential, high voltage pulsed current and neuromuscular waveforms in sequence. The device runs continuously for the first 2 days following surgery, then runs 3 times a day for 1 hour on days 3 through 42.
  Arms: 2
Device: SurgiStim3 — The placebo device is programmed to run for the same amount of time, at the same schedule, using the same waveforms as the functional device over the course of the 42 days. The placebo device, however, will only increase to 80% of the patient-set amplitude after a one minute set-up period and will only turn on for 6 seconds of every minute (3s ramp up, 1s on time, 2s ramp down).
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether a functional electrical stimulation device, the SurgiStim3, decreases pain, pain medications and/or edema in patients undergoing anterior cruciate ligament repair.

ELIGIBILITY:
Inclusion Criteria:

* Agree to provide informed consent to be included within this ACL study
* Demonstrate a continued willingness to be compliant with the parameters established under the study;
* Have no history of drug or alcohol abuse in the last 2 years;
* Be either a male or female adult between the ages of 18 and 64;
* Be undergoing a surgical repair of the anterior cruciate ligament (ACL) using either a hamstring, patella tendon, Achilles tendon, or allograft procedure; and
* Understand that there is no financial remuneration for participation in the study.

Exclusion Criteria:

* Pregnant women
* Insulin dependent diabetic patients
* Patients with a demand type pacemaker
* Patients who have a malignant tumor (other than basal cell epithelioma)
* Patients with a known history of alcohol or drug abuse in the last 2 years
* Patients who will not agree to provide informed consent to be included within this ACL study
* Patients who demonstrate a continued unwillingness to be compliant with the parameters established under this study.
* "Poor healers" as identified by the patient's medical history
* Patients who have a history of sensitivity to surgical tape, electrode adhesives, etc.
* Patients with a known history of RSD (reflex sympathetic dystrophy)
* Patients with a history of chronic pain (on opiates or high dosage of NSAIDS for 3 months or greater)
* Patients who have previously undergone an ACL reconstruction on the same knee
* Patients with clinically varicose veins (clinically significant or symptomatic)
* Patients whose history shows an abuse of diuretics or anti-inflammatory medications
* Patients who will undergo multiple ligament surgery (i.e., ACL plus PCL, MCL, and/or LCL)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
pain | post-op days 1, 3, 5, 7, 14, 21, 28, 35, 42

SECONDARY OUTCOMES:
pain medications | post-op days 1, 3, 5, 7, 14, 21, 28, 35, 42
edema | post-op days 7, 14, 21, 28, 35, 42

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Getelman, MD, Principal Investigator — Southern California Orthopedic Institute
Locations (1):
- Southern California Orthopedic Institute, Van Nuys, California, United States